CLINICAL TRIAL: NCT07216599
Title: Photoacoustic Imaging in Wound Evaluation and Treatment Guidance
Brief Title: Photoacoustic Imaging of Foot Wound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Jun Xia, Ph.D., Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009530; 5R01EB028978-04 (NIH)
Record Dates: First submitted 2025-10-02; First posted 2025-10-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Foot Ulcer
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single study arm (Experimental): Participants will undergo imaging using the investigational photoacoustic device.
  Interventions: Device: Photoacoustic imaging and multispectral imaging

INTERVENTIONS:
Device: Photoacoustic imaging and multispectral imaging — Use photoacoustic and Kent imaging devices that can image vasculature and assess tissue perfusion on the foot.

SUMMARY:
This pilot device trial aims to test the feasibility of using photoacoustic images to monitor tissue perfusion and to guide post-surgical wound treatment. Through this pilot study, the investigators will test the feasibility, identify any practical issues, and acquire essential information (e.g., drop-off rate, variation in wound healing rate) to guide future large-scale studies.

DETAILED DESCRIPTION:
This pilot device trial aims to test the feasibility of using photoacoustic images to monitor tissue perfusion and to guide post-surgical wound treatment. Through this pilot study, the investigators will test the feasibility, identify any practical issues, and acquire essential information (e.g., drop-off rate, variation in wound healing rate) to guide future large scale studies.

For recruited patients, wound care will be guided by both photoacoustic imaging and Kent imaging, a multi-spectral imaging technique for tissue oxygenation mapping. None of the techniques is currently used in the clinic as standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a chronic wound on the foot that is presumed to be due to arterial insufficiency.

Exclusion Criteria:

* Patients with a massive deep tissue infection.
* Patients with preexisting skin conditions, such as melanoma, psoriasis, in areas close to the wound(s).
* Noncompliant patients who do not adhere to care plans.
* Pregnant women.
* Adults unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment fidelity rate | 12 months
  The ratio of cases received additional clinical assessment due to photoacoustic imaging results.
Percentile healing score | 12 months
  The healing score will be defined as the ratio of the healed wound area versus the pre-treatment wound area (1-(post-treatment wound area)/(pre-treatment wound area)). A percentile healing value of 100% indicates that the wound is fully healed, while a value of 0% indicates that the wound area does not change.

SECONDARY OUTCOMES:
Recruitment rate | 12 months
  The ratio of recruited patients to the total number of eligible patients

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Vascular Surgery, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided